CLINICAL TRIAL: NCT06425445
Title: Development of a New Clinical Tool for the Assessment of Orofacial Muscles in Patients Affected by Facioscapulohumeral Muscular Dystrophy: a Preliminary Study.
Brief Title: Quantitative Assessment of Orofacial Muscle Function in FSHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mons (Other)
Responsible Party: Principal Investigator, Alexandre Legrand, Professor and Dean of the Faculty of Medicine and Pharmacy, University of Mons
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P2024/031
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Affected participants (Experimental)
  Interventions: Procedure: Measurement of maximal expiratory pressures during forced static expiratory maneuvers sustained over 5 seconds
- Healthy participants (Experimental)
  Interventions: Procedure: Measurement of maximal expiratory pressures during forced static expiratory maneuvers sustained over 5 seconds

INTERVENTIONS:
Procedure: Measurement of maximal expiratory pressures during forced static expiratory maneuvers sustained over 5 seconds — Participants perform forced static expiratory maneuvers sustained over a five second period

SUMMARY:
The goal of this study is to validate a new method for the assessment of orofacial muscles in FSHD affected individuals, using maximal expiratory pressures (MEPs).

Our hypothesis is the following:

- The pressure drop observed when using circular mouthpieces (versus ovoid mouthpieces) is a reflection of orofacial dysfunction in FSHD affected individuals

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of FSHD type 1 and/or type 2

Exclusion Criteria:

* Pregnant women
* Presence of other associated neuromuscular conditions
* Any unstable interfering clinical situation

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
The pressure drop | The pressure drop will be assessed for each study participant at visit 1 and subsequently at visit 2 (3 months later). The measurements as such, should take about 30 minutes for each participant
  The pressure drop (PD) is defined as the pressure difference between a reference ovoid-shaped mouthpiece and variously-sized circular mouthpieces, divided by the reference pressure. It is a relative value that is expected to reflect the magnitude of orofacial muscle dysfunction in FSHD affected individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Legrand (PhD, MD, principal investigator), Principal Investigator — University of Mons
Locations (1):
- University of Mons, Mons, Hainaut, Belgium